CLINICAL TRIAL: NCT04365816
Title: Evaluation of the Repercussions of the Coronavirus (Covid 19) Infection on Nutritional Health Status and Nutritional Care : an Observational French Cohort Study One Month After Their Discharge From Hospital
Brief Title: NutriCovid30 : Nutritional Evaluation for Covid-19 Infection at D30
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Grenoble Alps (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A01120-39
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Prospective cohort University Hospital, Grenoble: Semi-structured survey administered on the phone, once, one month after discharge from hospital. The interview will not be recorded.
  Interventions: Other: Interview
- Prospective cohort University Hospital, Toulouse: Semi-structured survey administered on the phone, once, one month after discharge from hospital. The interview will not be recorded.
  Interventions: Other: Interview
- Prospective cohort University Hospital, Nancy: Semi-structured survey administered on the phone, once, one month after discharge from hospital. The interview will not be recorded.
  Interventions: Other: Interview
- Prospective cohort University Hospital, Rennes: Semi-structured survey administered on the phone, once, one month after discharge from hospital. The interview will not be recorded.
  Interventions: Other: Interview
- Prospective cohort Hospices Civils de Lyon: Semi-structured survey administered on the phone, once, one month after discharge from hospital. The interview will not be recorded.
  Interventions: Other: Interview
- Prospective cohort Assistance Publique Hôpitaux de Paris: Semi-structured survey administered on the phone, once, one month after discharge from hospital. The interview will not be recorded.
  Interventions: Other: Interview
- Prospective cohort University Hospital, Rouen: Semi-structured survey administered on the phone, once, one month after discharge from hospital. The interview will not be recorded.
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — A survey was created, aiming to collect information about prior history of chronic disease, the Self-Evaluation of Food Intake, dysregulations (anosmia, ageusia...), anthropometric data, food data during and after hospitalisation, healthcare consumption since the discharge from hospital

SUMMARY:
Describe the main clinical features impacting the food intake, and therefore the nutritional status of a population infected by a coronavirus.

DETAILED DESCRIPTION:
The recent Covid-19 outbreak has brought USA, European, British and French nutrition learned societies to publish recommendations for the nutritional management of patients infected with the SARS-CoV-2. They reminded that there is a risk of malnutrition for that population.

The emergency and rapid evolution in the situation have led to severe cases of anosmia, ageusia, diarrhea, odynophagia, anorexia etc.. Some of the first patients cured from Covid-19 have lost up to 10 kgs.

To this day, there is no available information regarding either nutritional characteristics or nutritional interventions (enteral or parenteral nutrition, oral nutritional supplements, dietary supplementations) for Covid-19 patients.

The objective of this study is to describe nutritional consequences of the Covid-19 infection for adults, 30 days after their discharge from hospital, as well as the nutritional care they received.

Type and proportion of chronic diseases will be assessed in this trial.

ELIGIBILITY:
Inclusion Criteria:

* 30 days or more after discharge from hospital for Covid-19
* Patient received information about the trial and gave his/her consent
* Patient capable of answering the phone (alone or with some help)

Exclusion Criteria:

* Patient diseased
* impossibility to collect information from the patient or one of his/her relatives
* Patient protected by the French Public Health Code (art. L1121-5 à L1121-8)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited after they are discharged from Hospital Covid Units
Sampling Method: Non-Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of food intake at 1 month after discharge from hospital for COVID | one month after hospital discharge
  Self assessment on the SEFI (Self-Evaluation of Food Intake) scale at one month after hospital discharge: 0 corresponds to the worsen score (no ingesta) and 10 corresponds to the best (same ingesta than before the disease)

SECONDARY OUTCOMES:
Weight variation during the infection | one month after hospital discharge
  Self-reported weight in kilograms, or in the absence of self-reported variations before the disease, during hospitalisation, at hospital discharge, one month after hospital discharge
Clinical signs limiting food intake | one month after hospital discharge
  Effect of these factors (anorexia, dysgeusia, Ear Nose and Throat pain, swallowing disorders, intestinal transit disorders...) on SEFI and weight
Factors limiting food intake | one month after hospital discharge
  Effect of these factors (supply difficulties, disease-related food disgust, limiting food habits or prior diet, hydration difficulties, need for help) on SEFI and weight
Implemented nutritional strategy | one month after hospital discharge
  Effect of nutritional strategy and interventions that were implemented (nutritional advice, adapted meals, oral nutritional supplementation, enteral and parenteral nutrition during hospitalisation and one month after hospital discharge) on SEFI and weight
Pre-existing chronic disorders | one month after hospital discharge
  Effect of pre-existing chronic disorders (pulmonary, chronic inflammatory bowel disease, cardio-vascular disease, diabetes, obesity, cognitive disorders, immunodepression, cancer, inflammatory joint disorder) on SEFI and weight
Covid-19 repercussions | one month after hospital discharge
  Quantifying unscheduled consultations or hospitalisations in the month following discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Marie-France VAILLANT, PhD, Principal Investigator — Centre Hospitalier Universitaire Grenoble Alpes
Locations (1):
- Marie-France VAILLANT, Grenoble, France

IPD SHARING:
Plan to Share IPD: No